CLINICAL TRIAL: NCT01315704
Title: Maladie d'Alzheimer et Maladies apparentées : Caractérisation Des Anomalies Cognitivo-motrices, et Des Effets Des médicaments Anti-démence et de la Vitamine D à Partir de la Mise en Place d'Une Base de données au CMRR du CHU d'Angers
Brief Title: Alzheimer's Disease and Related Disorders
Acronym: MERE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Cédric ANNWEILER ; MD, Memory Centre of Angers University Hospital
Other Study IDs: 2009-15
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer's Disease; Gait Apraxia; Impaired Cognition
MeSH Terms: conditions — Alzheimer Disease; Gait Apraxia; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Patients with Mild Cognitive Impairment
  Interventions: Drug: Drug intervention
- Group 2: Patients with Mild Alzheimer's disease or related disorders
  Interventions: Drug: Drug intervention
- Group 3: Patients with Moderate Alzheimer's disease or related disorders
  Interventions: Drug: Drug intervention

INTERVENTIONS:
Drug: Drug intervention — before-after interventional (anti-dementia drugs and/or vitamin D) study
  Other Names: Anti-dementia drugs and/or vitamin D

SUMMARY:
The purpose of this study is to compare characteristics of gait and balance measured among patients with Alzheimer's disease or related disorders separated into 3 groups according to the stage of disease (i.e., pre-dementia, mild and moderate dementia stages); to determine the effects of anti-dementia drugs and vitamin D on cognitive motor abnormalities; and to establish a database at Angers University Memory Centre.

DETAILED DESCRIPTION:
Although gait disorders are frequently associated with Alzheimer's disease and related disorders (ADRD), few studies have focused on cognitive motor effects of anti-dementia drugs and vitamin D.

The objectives of this study are to

* Compare characteristics of gait and balance measured among patients with ADRD separated into 3 groups according to stages of disease (i.e., pre-dementia, mild and moderate dementia stages)
* To determine the effects of anti-dementia drugs and vitamin D on cognitive motor abnormalities
* To determine whether motor abnormalities could be associated with cognitive impairments, specifically executive dysfunctions
* To establish a database at Angers University Memory Center.

ELIGIBILITY:
Inclusion Criteria:

* All elderly patients from the University Memory Center of Angers University Hospital.
* Able to walk without any walking aid on 15 meters
* Mini-Mental Status Examination score > 10
* Being affiliated to a social security regime

Exclusion Criteria:

* Mini-Mental Status Examination score ≤ 10
* Subject suffering from pre-existing impellent disturbances
* History of cerebrovascular accident or other cerebro-spinal pathology
* Poor workmanship of the written or oral French language
* Use of walking aid such as walking frame with wheels or tricycle.
* Acute medical or surgical disease in the past 3 months
* Refusal to participate (or trustworthy person)
* Near visual acuity < 2/10

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients of the University Memory Center of Angers University Hospital with respect to the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2009-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Spatiotemporal gait parameters | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cedric ANNWEILER, MD, Principal Investigator — Memory Centre of Angers University Hospital
Locations (1):
- Cédric ANNWEILER , MD, Angers, France

REFERENCES:
- [Derived] Beauchet O, Barden J, Liu-Ambrose T, Chester VL, Annweiler C, Szturm T, Grenier S, Leonard G, Bherer L, Allali G; Canadian Gait Consortium. Anti-Dementia Drugs, Gait Performance and Mental Imagery of Gait: A Non-Randomized Open-Label Trial. Drugs Aging. 2016 Sep;33(9):665-73. doi: 10.1007/s40266-016-0391-0. PMID 27568453
- [Derived] Beauchet O, Launay CP, Allali G, Watfa G, Gallouj K, Herrmann FR, Annweiler C. Anti-dementia drugs and changes in gait: a pre-post quasi-experimental pilot study. BMC Neurol. 2013 Nov 21;13:184. doi: 10.1186/1471-2377-13-184. PMID 24261605